CLINICAL TRIAL: NCT04340804
Title: Socioeconomic Position and the Effect of kcal Labelling and PACE Labelling on Self-served Portion Size
Brief Title: Effect of kcal and PACE Labelling on Self-served Portion Size
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Responsible Party: Principal Investigator, Eric Robinson, Principal Investigator, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 803194 1B4
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Diet, Healthy; Food Selection
Keywords: kcal labelling; PACE labelling; portion size; socio-economic position
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Kcal labelling (Experimental): Participants allocated to this group will see on the screen the amount of food increasing or decreasing based on how many times they tap on the corresponding keys and a real-time kcal counter synchronised with the food amount changes (i.e., increasing/decreasing).
  Interventions: Behavioral: Kcal labelling
- PACE labelling (Experimental): Participants allocated to this group will see on the screen the amount of food increasing or decreasing based on how many times they tap on the corresponding keys and a real-time PACE counter (as minutes needed to walk to burn off the calories) synchronised to the food amount changes (i.e., increasing/decreasing) with 4 min being equivalent to 20 kcal.
  Interventions: Behavioral: PACE labelling
- Kcal and PACE labelling (Experimental): Participants allocated to this group will see on the screen the amount of food increasing or decreasing based on how many times they tap on the corresponding keys and a real-time kcal and PACE counters synchronised to the food amount changes (i.e., increasing/decreasing).
  Interventions: Behavioral: Kcal labelling; Behavioral: PACE labelling
- No labelling (No Intervention): Participants allocated to this group will only see on the screen the amount of food increasing or decreasing based how many times they tap on the corresponding keys.

INTERVENTIONS:
Behavioral: Kcal labelling — Real-time kcal counter synchronised with the food amount changes
  Arms: Kcal and PACE labelling; Kcal labelling
Behavioral: PACE labelling — Real-time PACE counter (as minutes needed to walk to burn off the calories) synchronised to the food amount changes
  Arms: Kcal and PACE labelling; PACE labelling

SUMMARY:
Participants will take part in an online survey. They will be asked to choose the amount of food they would like to eat based on pictures of 18 dishes sequentially displayed on the screen. They will be randomly allocated to four different groups: kcal labelling, PACE labelling (Physical Activity Calorie Equivalent: minutes to walk to burn off the calories), kcal and PACE labelling combined, no labelling, in a between subject design. The main outcome variable is the total "self-served" energy for each dish (in kcal).

DETAILED DESCRIPTION:
See attached protocol documents.

ELIGIBILITY:
Inclusion Criteria:

* United Kingdom residents
* Age ≥ 18
* Fluent in English
* Have access to a computer and Internet

Exclusion Criteria:

* Have any dietary restriction (vegetarian, vegan, gluten-free, sugar-free, diary or lactose free, food allergy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-05-13 (Actual)

PRIMARY OUTCOMES:
Total self-served energy (kcal) | 10 minutes (the time frame denotes time taken to perform the portion selection task and there is no follow up)
  Energy content of the portion selected for each dish.

SECONDARY OUTCOMES:
Kcal influence | 3 minutes (the time frame denotes time taken to fill in the debriefing questionnaire and there is no follow up)
  Whether kcal content influences the quantity of self-served food
PACE influence | 3 minutes (the time frame denotes time taken to fill in the debriefing questionnaire and there is no follow up)
  Whether physical activity energy equivalent influences the quantity of self-served food.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liverpool, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Shared on the Open Science Framework
Supporting Information: Study Protocol, SAP, ICF
Time Frame: On publication, indefinitely
Access Criteria: Open website
URL: https://osf.io/k369t/

REFERENCES:
- Available data/document: Study Protocol — https://osf.io/k369t/
- Available data/document: Statistical Analysis Plan — https://osf.io/k369t/
- Available data/document: Informed Consent Form — https://osf.io/k369t/
- Available data/document: Individual Participant Data Set — https://osf.io/k369t/ — When results will be published

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/04/NCT04340804/Prot_SAP_ICF_000.pdf